CLINICAL TRIAL: NCT07005284
Title: A Single-Ascending Dose Study to Evaluate the Safety and Pharmacokinetics of LY3981314 in Healthy Participants
Brief Title: A Study of LY3981314 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27406; J6H-MC-KXAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-06-03; First posted 2025-06-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3981314 Part A (Experimental): Single-ascending doses of LY3981314 administered subcutaneously (SC)
  Interventions: Drug: LY3981314
- LY3981314 Part B (Experimental): Single dose of LY3981314 administered SC
  Interventions: Drug: LY3981314
- Placebo Part A (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- Placebo Part B (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3981314 — Administered SC
  Arms: LY3981314 Part A; LY3981314 Part B
Drug: Placebo — Administered SC
  Arms: Placebo Part A; Placebo Part B

SUMMARY:
The main purpose of this study is to investigate the safety of LY3981314 when administered subcutaneously (SC) (under the skin), and how it's processed in the body.

The study will last approximately 25 weeks, excluding a screening period with an optional extension to approximately 49 weeks for qualifying participants.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and 12-lead electrocardiogram (ECG)
* Individuals assigned male at birth who agree to follow contraceptive requirements, or individuals assigned female at birth and not of childbearing potential
* Have venous access sufficient to allow for blood sampling
* Have a body weight within 45 to 145 kilograms (kg) and body mass index within the range of 18.5 to 35 kilogram per square meter (kg/m²) (inclusive)
* For Part B:

  * Japanese participants must be first-generation Japanese, defined as the participant, the participant's biological parents, and all of the participant's biological grandparents being of exclusive Japanese descent and born in Japan
  * To qualify as Chinese for this study, all 4 of the participant's biological grandparents must be of exclusive Chinese descent and born in China

Exclusion Criteria:

* Have known allergies to LY3981314, related compounds, or any components of the formulation
* Have a significant history of or current rheumatologic, cardiovascular, respiratory, renal, gastrointestinal, endocrine (such as Cushing syndrome, hyperaldosteronism), hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational medicinal product; or of interfering with the interpretation of data
* Have received at least 1 live vaccine within 28 days of screening, or intend to do so during the study, or within 28 days after the study
* Had any surgical procedure (except for minor surgery requiring local or no anesthesia and without any complications or sequelae) within 12 weeks prior to screening, or intend to do so during the study, or within 28 days after the study
* Show evidence of active or latent tuberculosis (TB)
* Have used, or intend to use, prescription or nonprescription medication within 14 days prior to dosing (or 5 half-lives - whichever is longer)
* Have a diagnosis or history of malignant disease
* Have a history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the participant to infection that, in the opinion of the sponsor or investigator, poses an unacceptable risk to the participant
* Have had any significant infections within 3 months prior to the screening visit or develop any of these infections before the randomization visit
* Have used, or intend to use, prescription or nonprescription medication within 14 days prior to dosing (or 5 half-lives - whichever is longer)
* Have participated in a clinical study involving an investigational product within the last 30 days of the final drug administration (or 5 half-lives, whichever is longer)
* Have donated 500 milliliters (mL) of blood or more or participated in a clinical study that required a blood volume of at least 500 mL, within the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Approximately Week 25
  A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3981314 | Baseline Up to Approximately Week 25
  PK: AUC of LY3981314
PK: Maximum Concentration (Cmax) of LY3981314 | Baseline up to Approximately Week 25
  PK: Cmax of LY3981314

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- CenExel ACT, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No